CLINICAL TRIAL: NCT07378839
Title: Alternate Nostril Breathing (ANB) for 1st Trimester Nausea and Vomiting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBGYN-2025-34216
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Emesis; Nausea
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate Nostril Breathing (Active Comparator): Participants in the intervention group will receive a brief orientation via a research team member at the time of randomization on alternate nostril breathing (ANB) and then be provided with a written and video-based instructional guide. They will be instructed to perform ANB 3 times per day for 5-10 minutes per session over a 7-day period and document their sessions in a daily symptom diary. The 7-day period will begin the following day after enrollment to allow for a full day of intervention implementation (Day 1-7).
  Interventions: Behavioral: Alternate Nostril Breathing
- Usual Care Only (No Intervention): This group will receive usual care and complete a daily symptom diary for Day 1-7.

INTERVENTIONS:
Behavioral: Alternate Nostril Breathing — ANB 3 times per day for 5-10 minutes per session over a 7-day period
  Arms: Alternate Nostril Breathing

SUMMARY:
This is a prospective, two-arm, non-blinded randomized controlled study designed to evaluate the effects of a one-week alternate nostril breathing (ANB) intervention on nausea and vomiting severity in pregnant individuals during their first trimester.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals aged 18 years or older
* Viable pregnancy with a gestational age between 6 0/7 - 12 6/7 weeks of gestation, confirmed by last menstrual period or ultrasound
* Diagnosed with mild to moderate NVP (PUQE-24 score between 4-12)
* Ability to understand and read English

Exclusion Criteria:

* Severe nausea and vomiting, defined as a PUQE score >12, or diagnosis of hyperemesis gravidarum requiring hospitalization or intravenous fluid therapy
* Pre-existing, active or acute respiratory conditions (e.g., asthma, COPD)
* History of severe anxiety disorders affecting breathing patterns
* Known deviated nasal septum
* Nausea and vomiting that pre-dates the pregnancy or is suspected to be due to a etiology other than pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Severity of Nausea and Vomiting | Day 7
  Measured by the change in the Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) score, where scores range from 3-15, and a higher score indicates greater severity of nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Babbar, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States